CLINICAL TRIAL: NCT05507320
Title: Neural Circuits for Action Perception
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Gabriel Kreiman, Professor, Boston Children's Hospital
Other Study IDs: IRB_P0405065R
Record Dates: First submitted 2022-08-09; First posted 2022-08-18 (Actual); Last update posted 2022-08-18 (Actual); Status verified 2022-08

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Mechanisms of action perception and execution — Study the mechanisms of action perception and execution

SUMMARY:
Study the mechanisms underlying action recognition and execution

DETAILED DESCRIPTION:
Subjects will participate in a task where they have to either

1. Perform a movement
2. Observe an actor performing a movement There are three types of actions including different kinematics and grip types The goal is to compare the neural circuits activated by action execution versus action observation.

ELIGIBILITY:
Inclusion Criteria:

* Patients with pharmacologically intractable epilepsy

Exclusion Criteria:

* Any situation that may put the patient at risk

Ages: 14 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with pharmacologically intractable epilepsy undergoing invasive implantation of electrodes
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Selectivity for kinematics and movement type in neurophysiological responses | Through study completion, an average of 2 years.
  Measure intracranial field potentials (in microvolts) in the gamma frequency band through neurophysiological responses comparing neural responses during action perception versus execution.
  We will assess selectivity for kinematics for each movement type
Evoked responses by action execution | Through study completion, an average of 2 years.
  Measure intracranial field potentials (in microvolts) in the gamma frequency band through neurophysiological responses comparing neural responses during action perception versus execution.
  We will quantify responses evoked by action execution
Evoked responses by action observation | Through study completion, an average of 2 years.
  Measure intracranial field potentials (in microvolts) in the gamma frequency band through neurophysiological responses comparing neural responses during action perception versus execution.
  We will quantify responses evoked by action observation

CONTACTS AND LOCATIONS:
Overall Officials: Gabriel Kreiman, PhD, Principal Investigator — CHB
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No